CLINICAL TRIAL: NCT00096642
Title: Comprehensive Treatment for Depressed Youth: An Outcome Evaluation Study
Brief Title: Cognitive Behavioral Therapy for Early-Onset Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Katharina Manassis, MD, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBT DEP; Ethics # 138/2001
Record Dates: First submitted 2004-11-12; First posted 2004-11-15 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Major Depressive Disorder; Dysthymic Disorder
Keywords: cognitive behavioral therapy; depression; group therapy; parenting; children and adolescents
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive behaviour versus standard care

SUMMARY:
Depression is a debilitating illness affecting large numbers of young people. In this study, children and adolescents ages 10 to 17 meeting criteria for clinical depression will participate in a 15-session group therapy (cognitive behavioral therapy or CBT) that teaches strategies for overcoming depressed mood. For half the participants, their parents will also participate in a parent group. By studying the role of parental involvement, we hope to develop more effective treatments for depressed children and teens in the future.

DETAILED DESCRIPTION:
Depression is a debilitating illness affecting large numbers of young people. Psychotherapy approaches have shown some promise in teens, but few studies have examined these interventions when offered in a group format. The role of parents in treatment outcome has also received little attention.

In this study, children and adolescents ages 10 to 17 meeting criteria for clinical depression will participate in a 15-session group therapy (cognitive behavioral therapy or CBT) that teaches strategies for overcoming depressed mood. For half the participants, their parents will also participate in a parent group to help them better manage their depressed children and teens. We will randomly assign children to CBT with or without parental involvement. We hope to show that involving parents results in additional improvements in the children. We will also study factors that predict which children do best in treatment, and maintenance of gains at 6 month and 1 year follow-up. These findings will allow us to provide more effective treatments to depressed children and teens in the future.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents meeting DSM-IV criteria for either Major Depression or Dysthymic Disorder.

Exclusion Criteria:

* Psychotic,
* Actively suicidal,
* IQ less than 80,
* Unable to speak English

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2002-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Diagnosis on structured interview | pre and post-intervention
Children's Depression Inventory score | pre- and post-intervention

SECONDARY OUTCOMES:
Multidimensional Anxiety Scale for Children | pre- and post-intervention
Children's Global Assessment Scale | pre- and post-intervention
Brief Family Assessment Measure | pre- and post-intervention
Perceived Competence Scale for Children | pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Manassis, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Birmaher B, Ryan ND, Williamson DE, Brent DA, Kaufman J, Dahl RE, Perel J, Nelson B. Childhood and adolescent depression: a review of the past 10 years. Part I. J Am Acad Child Adolesc Psychiatry. 1996 Nov;35(11):1427-39. doi: 10.1097/00004583-199611000-00011. PMID 8936909
- [Background] Birmaher B, Ryan ND, Williamson DE, Brent DA, Kaufman J. Childhood and adolescent depression: a review of the past 10 years. Part II. J Am Acad Child Adolesc Psychiatry. 1996 Dec;35(12):1575-83. doi: 10.1097/00004583-199612000-00008. PMID 8973063
- [Background] Birmaher B, Brent DA, Kolko D, Baugher M, Bridge J, Holder D, Iyengar S, Ulloa RE. Clinical outcome after short-term psychotherapy for adolescents with major depressive disorder. Arch Gen Psychiatry. 2000 Jan;57(1):29-36. doi: 10.1001/archpsyc.57.1.29. PMID 10632230
- See also: Website of American Academy of Child & Adolescent Psychiatry — http://www.aacap.org